CLINICAL TRIAL: NCT05671016
Title: Brain Imaging to Predict Toxicity in Elderly Patients After Radiotherapy
Acronym: BRITER
Status: Completed | Type: Observational
Sponsor: Brighton and Sussex University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: BRITER
Record Dates: First submitted 2022-11-29; First posted 2023-01-04 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2022-12

CONDITIONS: Glioblastoma Multiforme, Adult; Radiation Toxicity; Quality of Life
MeSH Terms: conditions — Glioblastoma; Radiation Injuries | interventions — Magnetic Resonance Spectroscopy; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient aged 65 or older receiving radiotherapy treatment for a newly diagnosed GBM: Patients aged 65 or older who have been newly diagnosed with a Glioblastoma (either through histological confirmation or confirmed by a consultant radiologist in a multidisciplinary team meeting setting) who are planned to be treated with radiotherapy. There is only 1 arm in this study, there is no randomisation. All participants will undertake questionnaires (as described in detail elsewhere in the form) and if the required MRI sequences are not available on their diagnostic imaging then they will undertake a trail specific MRI scan.
  Interventions: Procedure: MRI scans and questionnaires

INTERVENTIONS:
Procedure: MRI scans and questionnaires — Extra baseline MRI scan performed and questionnaires (EORTC validated questionnaires involving EORTC QLQ C-30, EORTC BN20 and EORTC ELD14) to assess quality of life at baseline, 4 weeks and 8 weeks after treatment

SUMMARY:
The investigators' aim with the BRITER study is to produce a way of predicting who might be more or less likely to suffer side effects from radiotherapy prior to starting treatment for a glioblastoma (GBM), a type of brain tumour.

GBM is the commonest primary malignant brain tumour. Treatment options include chemotherapy, radiotherapy or best supportive care. The focus should be on maintaining a good quality of life for as long as possible.

Radiotherapy to the brain is an effective treatment, however it can produce side effects. The degree of side effects different patients experience can vary widely. It has been thought that if the patient's underlying normal brain is fragile due to an underlying mild dementia or problems associated with high blood pressure or cholesterol then this might make them more vulnerable to radiotherapy.

MRI scans can be used to assess whether there are changes in the normal brain. The BRITER study aims to use MRI scans to see whether the investigators can predict those patients who might be more at risk of side effects from radiotherapy. The trial is aimed at patients aged > 65 who have been newly diagnosed with a GBM and are going to receive radiotherapy. Patients who agree to take part in the trial will have had an MRI scan as part of their normal diagnosis. Participants will undertake some questionnaires before starting their radiotherapy which will aim to assess their quality of life and their mental processes of perception, memory, judgment, and reasoning (called cognitive function). Participants may also need an extra MRI scan.

Participants will repeat these questionnaires 4 and 8 weeks after treatment when they come for their follow up appointments. The investigators will compare them to measurements made on the pre-treatment MRI scan.

Participation in the study does not change the treatment the patient receives.

The investigators hope that the BRITER study will enable them to predict the degree of side effects a patient is likely to experience before embarking on radiotherapy treatment. This will enable more informative, individualised discussions surrounding the best treatment path for older patients with a GBM.

DETAILED DESCRIPTION:
Glioblastoma (GBM) is the commonest primary malignant brain tumour among the adult population with approximately 2,000 new cases diagnosed in the UK per year. Incidence peaks in the 7th and 8th decades of life and as the global population ages, rates are increasing. Outcomes from this disease remain poor with median life expectancy in the range of 12-18 months, dropping to 3-6 months in the older population. The reasons for this are multifactorial, including more aggressive tumour biology in the older age group, decreased tolerance to treatment related side effects and the potential of under treatment by doctors within the older age group.

Given the poor prognosis in this group, treatment must be balanced against side effects and worsening quality of life. In patients aged 65 or over there is a lack of consensus on standard of care. Radiotherapy has a survival advantage over best supportive care however the optimal dose of radiotherapy is yet to be established. A recent Phase III trial randomised elderly GBM patients to standard radiotherapy with 60Gy in 30#, hypofractionated radiotherapy of 34Gy in 10# or temozolomide (TMZ) chemotherapy alone. For patients older than 65, survival was significantly longer with TMZ or hypofractionated radiotherapy than with standard radiotherapy . Those with defects in the DNA repair protein MGMT did significantly better in the chemotherapy arm than those with intact MGMT, a result which was replicated in the NOA-08 trial which randomised elderly GBM patients to standard radiotherapy with 60Gy in 30# or TMZ alone. This non-inferiority trial showed TMZ to be a suitable monotherapy option, with greater effect seen in those with MGMT promoter methylation . Recently published evidence has shown a survival benefit from adding concomitant and adjuvant TMZ to a hypofractionated radiotherapy regime of 40Gy in 15# in patients aged over 65, again with greater effect seen in those with MGMT promoter methylation . There is therefore now evidence to support the use of concomitant chemoradiotherapy or chemotherapy or radiotherapy as single agents amongst elderly GBM patients and an increasing interest in using MGMT promoter methylation status as a biomarker. However there remains a paucity of data surrounding the clinical and radiological basis by which individual patients are assessed for treatment.

The majority of GBM patients over 65 who are actively treated by oncologists receive some form of radiotherapy to the brain. Short term side effects from radiotherapy include fatigue, headache, cognitive defects, nausea, weakness and a need for increased steroid doses. Longer term side effects include persistent cognitive defects, long term fatigue and hormonal imbalances . Radiation causes an inflammatory response within the brain tissue as well as disrupting the blood brain barrier. It affects the vasculature of the brain with endothelial cell damage leading to microvascular dilatation, thickening of the vessel wall and increased risk of microbleeds and ischemic strokes in the months to follow . There is a risk of inducing tissue necrosis from occlusion of small blood vessels within the brain parenchyma, leading to coagulation, focal necrosis and demyelination. Animal models have suggested radiation is cytotoxic to developing neuroglial progenitor cells with areas of stem cells such as the hippocampus and periventricular zones, particularly vulnerable to damage, leading to longer term neurocognitive decline . There is evidence to suggest that radiotherapy can stabilise or improve functional ability for some older patients with GBM as well as providing a survival advantage however clinical experience shows that the degree of side effects experienced and their impact on quality of life varies widely within this patient cohort.

Risk factors for toxicities from radiotherapy include dose, fractionation and age however there are no more accurate ways of predicting which patients are more likely to suffer side effects. MRI has been shown to accurately pick up microhaemorrhages and other ischemic changes which may correlate with a 'vulnerable' brain pre-treatment . These MRI changes have been examined in Alzheimer and dementia research with correlations shown between MRI markers and disease severity , however they have not yet been used within the neuro oncology setting.

The investigators aim to examine the relationship between MRI markers of a 'vulnerable' brain and degree of acute side effects and change in quality of life amongst a population of older patients being treated with cranial radiotherapy for GBM.

The poor prognosis of older GBM patients leads to an emphasis on the need for focusing on quality of life when deciding on treatment regimes. There are pathological markers which can help them determine the sensitivity of the tumour to chemotherapy however there is no such guidance when it comes to making decisions about radiotherapy. If it were possible to predict the degree of side effects likely to be experienced by a patient from radiotherapy treatment then it would enable clinicians to make more individually tailored, patient centred treatment plans.

The investigators aim to see if analysis of pre-radiotherapy MRI scans including T2 gradient echo and susceptibility weighted imaging sequences can correlate with acute treatment related toxicity and quality of life amongst patients aged 65 or over undergoing partial brain radiotherapy for GBM. As these patients have an average life expectancy of 3-6 months within the UK the investigators are focussing on acute rather than long term side effects of radiotherapy.

MRI sequences will be utilised to determine any markers of background subclinical microvascular or degenerative disease in the normal brain including microhaemorrhage secondary to hypertension or cerebral amyloid angiopathy and atrophy with cortical volume measurement of the contralateral hemisphere. Additional susceptibility weighted sequences will be performed to identify the presence of microhaemorrhages in the contralateral normal-appearing brain parenchyma. These will be semi-quantitatively assessed using a modified established microhaemorrhage scoring methodology. Absolute measures of the contralateral normal-appearing hemisphere cortical volumes will be acquired using FSL freesurfer software and a volumetric T1 weighted acquisition. These techniques will give the investigators a number of quantitative scores that can then assessed for correlation with changes in quality of life and toxicity scoring systems.

Radiotherapy is an effective palliative treatment for GBMs and has been shown in clinical trials to maintain or improve health related quality of life. However outside of a clinical trial population, usual clinical practice reveals some patients in whom the side effect profile from cranial radiotherapy is intolerable and has a significant detrimental effect on patients' quality of life for their remaining short lifespan. The BRITER study aims to examine whether analysis of pre-treatment MRI scans in this cohort could help to predict who is more vulnerable to these side effects and therefore reveal a group of patients in whom single agent chemotherapy or best supportive care would be better treatment options.

The BRITER study is being performed in patients aged 65 or over who have a new diagnosis of GBM. It tests the hypothesis that there is a relationship between 6 scores of a 'vulnerable' brain seen on pre-treatment MRI and a clinically significant change in patient quality of life, as defined by a 10 point change in the EORTC QLQ C30 questionnaire from baseline to 8 weeks post treatment.

ELIGIBILITY:
Inclusion Criteria:

* • Patients aged > 65 years with a new diagnosis of GBM. Diagnosis made via histological confirmation following biopsy or debulking surgery or radiologically during a Multidisciplinary meeting (MDM) confirmed by a consultant neuro radiologist. This lower age limit is due to previous clinical trials which have established gold standard treatment regimes for patients under the age of 65. Patients aged 65 or over have less clinical trial data available to them and treatment decisions are more nuanced with a greater emphasis on quality of life given the poorer prognosis of older patients.

  * Patients undergoing radiotherapy treatment to the brain for treatment of their GBM
  * Patients able to undergo an MRI scan
  * Patients undergoing treatment at one of the study centres
  * Patient have capacity to participate in the study
  * Patients with physical impairments that prevent them filling in their questionnaires involved in the study may still participate if they are able to communicate their answers though a third party

Exclusion Criteria:

* • Patients not fit for radiotherapy treatment or having single agent chemotherapy with no radiotherapy

  * Patients lacking capacity
  * Patients who do not have sufficient grasp of the English language to be able to complete the questionnaires
  * Patients unable to communicate their responses to the questionnaires
  * Patients who are concurrently enrolled in a Clinical Trial of an Investigational Medicinal Product (CTIMP)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients aged 65 or over with newly diagnosed Glioblastoma Multiforme planning to receive radiotherapy to the brain
Sampling Method: Non-Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Quality of Life at 8 weeks post treatment. | 8 weeks (+/- 1 week) after completing radiotherapy to the brain
  Participants will complete validated quality of life questionnaires at baseline and at 8 weeks after treatment. The main outcome measure is the EORTC QLQ-C30 questionnaire. This will be scored and then assessed for differences between baseline and the 8 week score to assess for a clinically significant (10 point change) in score. The scores shall be calculated using the EORTC scoring manual which involves reverse scoring some domains. A higher overall score indicates a better quality of life.

SECONDARY OUTCOMES:
Overall survival | This will be calculated from the date of diagnosis of a Glioblastoma to the date of death or the date the study is censored (set at 31/12/2021, 16 months after the final patient is recruited) whichever is first
  As calculated below
Change in score on MOCA cognitive screening questionnaire | at 8 weeks (+/- 1 week) after treatment complete
  The Montreal Cognitive Assessment is a cognitive screening test which is scored out of 30. A higher test score indicates better cognitive functioning. A score of 26 or below indicates impaired functioning. We will assess scores at baseline and at 8 weeks after treatment to check for changes in cognitive functioning
Change in score in EORTC BN20 questionnaire | Between baseline and 8 weeks
  The EORTC BN20 is a quality of life score specifically focussing on Brain related symptoms. It will be scored (higher score indicating better QoL) using the EORTC scoring manual. A linear model will be used
Change in score in EORTC ELD-14 questionnaire | Between baseline and 8 weeks
  Quality of life questionnaire focusing on elderly symptoms. A higher score indicates better quality of life. This will be scored using the EORTC scoring manual. A linear model will be used

OTHER OUTCOMES:
Total brain volume (as a ratio of total intracranial volume to CSF) (mm3) | Baseline
  This is one of six MRI based imaging variables that will be calculated on the participants' baseline MRI scan. These six measures represent a numerical way to score a 'vulnerable' brain parenchyma and will be modelled against the change in quality of life scores
Contralateral medial temporal lobe volume (mm3) | Baseline
  This is one of six MRI based imaging variables that will be calculated on the participants' baseline MRI scan. These six measures represent a numerical way to score a 'vulnerable' brain parenchyma and will be modelled against the change in quality of life scores
Volume of T1 white matter hyperintensities in contralateral hemisphere (mm3) | Baseline
  This is one of six MRI based imaging variables that will be calculated on the participants' baseline MRI scan. These six measures represent a numerical way to score a 'vulnerable' brain parenchyma and will be modelled against the change in quality of life scores
Number of white matter microhaemorrhages seen on T2* or SWI in contralateral hemisphere (range 0 to 7) | Baseline
  This is one of six MRI based imaging variables that will be calculated on the participants' baseline MRI scan. These six measures represent a numerical way to score a 'vulnerable' brain parenchyma and will be modelled against the change in quality of life scores
Fazakas scale assessing white matter changes on T2 weighted imaging calculated in contralateral hemisphere (range 0-3) | Baseline
  This is one of six MRI based imaging variables that will be calculated on the participants' baseline MRI scan. These six measures represent a numerical way to score a 'vulnerable' brain parenchyma and will be modelled against the change in quality of life scores
Radiotherapy planning target volume (cc) | Baseline
  This is one of six MRI based imaging variables that will be calculated on the participants' baseline MRI scan. These six measures represent a numerical way to score a 'vulnerable' brain parenchyma and will be modelled against the change in quality of life scores

CONTACTS AND LOCATIONS:
Overall Officials: Cressida Lorimer, MD, Study Chair — Brighton and Sussex NHS Trust
Locations (1):
- Scott Harfield, Brighton, Sussex, United Kingdom

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-04-03): https://cdn.clinicaltrials.gov/large-docs/16/NCT05671016/Prot_SAP_000.pdf
  • Informed Consent Form (2019-09-09): https://cdn.clinicaltrials.gov/large-docs/16/NCT05671016/ICF_001.pdf